CLINICAL TRIAL: NCT00936390
Title: A Phase III Prospective Randomized Trial of Dose-Escalated Radiotherapy With or Without Short-Term Androgen Deprivation Therapy for Patients With Intermediate-Risk Prostate Cancer
Brief Title: Radiation Therapy With or Without Androgen-Deprivation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0815; CDR0000648194; NCI-2011-01948 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Flutamide; Androgen Antagonists; Gonadotropin-Releasing Hormone; Therapeutics; Leuprolide; Goserelin; Buserelin; Triptorelin Pamoate; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose-Escalated Radiation Therapy Alone (Active Comparator): Radiation therapy consists of 79.2 Gy EBRT only or 45 Gy EBRT followed by low- or high-dose rate brachytherapy. EBRT is delivered in 1.8 Gy daily fractions.
  Interventions: Radiation: Dose-Escalated Radiation Therapy
- Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation (Experimental): Radiation therapy consists of 79.2 Gy EBRT only or 45 Gy EBRT followed by low- or high-dose rate brachytherapy. EBRT is delivered in 1.8 Gy daily fractions.
  Six months of androgen-deprivation therapy starts 8 weeks prior to start of radiation therapy and consists of luteinizing-hormone releasing-hormone (LHRH) agonist (antagonist) therapy (leuprolide, goserelin, buserelin. triptorelin, or degarelix) and anti-androgen therapy (bicalutamide or flutamide).
  Interventions: Drug: bicalutamide; Drug: flutamide; Drug: LHRH agonist (antagonist) therapy; Radiation: Dose-Escalated Radiation Therapy

INTERVENTIONS:
Drug: bicalutamide — Administered orally at a dose of one 50 mg tablet per day, beginning within (before, same day as, or after) 10 days of the date of the first LHRH agonist (antagonist) therapy administration and continuing for a total duration of 6 months.
  Arms: Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Drug: flutamide — Administered orally at a dose of 250 mg (two 125-mg capsules) three times a day for a total daily dose of 750 mg, beginning within (before, same day as, or after) 10 days of with the date of the first LHRH agonist (antagonist) therapy administration and continuing for a total duration of 6 months.
  Other Names: anti-androgen therapy
  Arms: Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Drug: LHRH agonist (antagonist) therapy — LHRH agonist (antagonist) therapy consists of leuprolide, goserelin, buserelin, triptorelin, or degarelix. The manufacturer's instructions should be followed. The first administration occurs with the start of anti-androgen treatment 8 weeks prior to the start of RT. The total duration of LHRH agonist (antagonist) therapy is 6 months.
  Other Names: leuprolide; goserelin; buserelin; triptorelin; degarelix
  Arms: Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Radiation: Dose-Escalated Radiation Therapy — External beam radiotherapy (EBRT) as 3D Conformal Radiotherapy (3DCRT) or intensity-modulated radiation therapy (IMRT). Brachytherapy is optional, at the discretion of the treating physician. Patients treated entirely via EBRT receive 79.2 Gy delivered in 1.8 Gy fractions. Patients who receive brachytherapy as a component of their RT receive 45 Gy EBRT in 1.8 Gy fractions. Low-dose brachytherapy boost occurs following the EBRT portion of treatment no more than 4 weeks following its completion.High-dose rate brachytherapy boost is delivered in 2 fractions separated by a minimum time span of 6 hours and the implant(s) may be performed during the EBRT portion of the treatment or within 1 week prior to its initiation or following its completion.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells and shrink tumors. Androgens can cause the growth of prostate cancer cells. Androgen-deprivation therapy may lessen the amount of androgens made by the body. It is not yet known whether radiation therapy is more effective with or without androgen-deprivation therapy in treating patients with prostate cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared with radiation therapy given together with androgen-deprivation therapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Demonstrate an overall survival (OS) advantage in patients with intermediate-risk prostate cancer treated with dose-escalated radiotherapy (RT) with versus without short-term androgen-deprivation therapy (ADT).

Secondary

* Determine whether the addition of ADT to dose-escalated RT versus RT alone improves clinical failures, biochemical failure by the "nadir +2", freedom from failure, rate of salvage ADT, and prostate cancer-specific mortality in these patients.
* Estimate the magnitude of benefit of ADT with respect to OS in patients treated with different RT modalities (i.e., external-beam radiation therapy alone vs low-dose rate brachytherapy boost vs high-dose rate brachytherapy boost).
* Compare acute and late treatment adverse events of these regimens and correlate these events with the presence or absence of pre-existing comorbidity as documented by the Adult Comorbidity Evaluation 27 assessment.

OUTLINE: This is a multicenter, dose-escalation study of radiotherapy. Patients are stratified according to number of risk factors (1 vs 2-3), comorbidity (ACE-27 grade ≥ 2 vs < 2), and radiotherapy (RT) modality (dose-escalated external-beam RT [EBRT] vs EBRT and low-dose rate brachytherapy boost vs EBRT and high-dose rate brachytherapy boost). Patients are randomized to 1 of 2 treatment arms. After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologically) proven diagnosis of prostatic adenocarcinoma, at intermediate risk for recurrence, within 180 days prior to registration as determined by having one or more of the following intermediate-risk features: Gleason score 7; prostate-specific antigen (PSA) >10 but ≤20; clinical stage T2b-T2c.

   * Patients previously diagnosed with low risk (Gleason score ≤ 6, clinical stage < T2a, and PSA < 10) prostate cancer undergoing active surveillance who are re-biopsied and found to have intermediate risk disease according to the protocol criteria are eligible for enrollment within 180 days of the repeat biopsy procedure.
2. Clinically negative lymph nodes as established by imaging (pelvic +/- abdominal CT or MRI), nodal sampling, or dissection within 60 days prior to registration, except as noted immediately below:

   * Patients with a single intermediate risk factor only do not require abdominopelvic imaging, but these studies may be obtained at the discretion of the treating physician. Patients with 2 or 3 risk factors are required to undergo pelvic +/- abdominal CT or MRI.
   * Patients with lymph nodes equivocal or questionable by imaging are eligible without biopsy if the nodes are ≤1.5 cm; any node larger than this on imaging will require negative biopsy for eligibility.
3. No evidence of bone metastases (M0) on bone scan within 60 days prior to registration.

   * Bone scan is not required for patients enrolled with a single intermediate risk factor only, but this scan may be obtained at the discretion of the treating physician. Patients with 2 or 3 risk factors will require a negative bone scan for eligibility.
   * Equivocal bone scan findings are allowed if plain film x-rays are negative for metastasis.
4. History/physical examination (to include, at a minimum, digital rectal examination of the prostate and examination of the skeletal system and abdomen, and formal comorbidity assessment via the ACE-27 instrument) within 60 days prior to registration.
5. Zubrod Performance Status 0-1
6. Age ≥ 18
7. Baseline serum PSA value performed with an FDA-approved assay (e.g., Abbott, Hybritech) within 60 days prior to registration

   * Study entry PSA must not be obtained during the following time frames: (1) 10-day period following prostate biopsy; (2) following initiation of ADT; (3) within 30 days after discontinuation of finasteride; or (4) within 90 days after discontinuation of dutasteride.
8. For patients undergoing brachytherapy only: complete blood count (CBC)/differential obtained within 60 days prior to registration, with adequate bone marrow function defined as follows:

   * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3
   * Platelets ≥ 100,000 cells/mm3
   * Hemoglobin (Hgb) ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
9. Patient must be able to provide study-specific informed consent prior to study entry.

Exclusion Criteria:

1. Patients with Gleason Score ≥ 8; PSA > 20; OR Clinical Stage ≥ T3 are ineligible for this trial.

   * Should findings of extracapsular extension or seminal vesicle invasion be noted on prostate MRI, this study, if used, will not render patients ineligible for accrual to this protocol. Primary tumor staging for eligibility purposes is to be based on palpable or core biopsy evidence only with respect to extracapsular extension or seminal vesicle involvement.
2. Patients with all three intermediate risk factors who also have ≥ 50% of the number of their biopsy cores positive for cancer are ineligible for this trial.
3. Prior invasive malignancy (except non-melanomatous skin cancer) or hematological (e.g., leukemia, lymphoma, myeloma) malignancy unless disease free for a minimum of 5 years (prior diagnoses of carcinoma in situ are permitted)
4. Prior radical surgery (prostatectomy), high-intensity focused ultrasound (HIFU) or cryosurgery for prostate cancer
5. Prior hormonal therapy, such as LHRH agonists (e.g., goserelin, leuprolide), antiandrogens (e.g., flutamide, bicalutamide), estrogens (e.g., DES), or bilateral orchiectomy
6. Use of finasteride within 30 days prior to registration
7. Use of dutasteride within 90 days prior to registration
8. Prior or concurrent cytotoxic chemotherapy for prostate cancer; prior chemotherapy for a different cancer is permitted.
9. Prior RT, including brachytherapy, to the region of the study cancer that would result in overlap of RT fields

   * Any patient undergoing brachytherapy must have transrectal ultrasound confirmation of prostate volume <60 cc, American Urological Association Symptom Index (AUA-SI) score ≤15 within 60 days of registration, and no history of prior transurethral resection of the prostate (TURP); prior TURP is permitted for patients who receive EBRT only)
10. Severe, active co-morbidity, defined as follows:

    * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
    * Transmural myocardial infarction within the last 6 months
    * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
    * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
    * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
    * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. While the treatment employed in this study is not significantly immunosuppressive, it is felt that a diagnosis of AIDS associated with prostate cancer is likely to impact this study's primary endpoint of overall survival. Patients who are HIV seropositive but do not meet criteria for diagnosis of AIDS are eligible for study participation.
11. Men who are sexually active with a woman of child-bearing potential and not willing/able to use medically acceptable forms of contraception (e.g., surgical, barrier, medicinal) during protocol treatment and during the first 3 months after cessation of protocol treatment; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1538 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro A. Martinez, MD, FACR, Study Chair — 21st Century Oncology - Michigan Institute for Radiation Oncology
Locations (518):
- United States (499):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - 21st Century Oncology-Scottsdale, Scottsdale, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - Mercy Cancer Center-Hot Springs, Hot Springs, Arkansas
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Enloe Medical Center, Chico, California
  - 21st Century Oncology - El Segundo, El Segundo, California
  - Fresno Cancer Center, Fresno, California
  - Saint Agnes Medical Center, Fresno, California
  - Marin General Hospital, Greenbrae, California
  - Veterans Administration Long Beach Medical Center, Long Beach, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Stanford Cancer Institute, Palo Alto, California
  - Feather River Cancer Center, Paradise, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - David Grant United States Air Force Medical Center, Travis Air Force Base, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - The Shaw Regional Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale-New Haven Hospital Saint Raphael Campus, New Haven, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - University of Miami Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Florida Hospital Kissimmee, Kissimmee, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - The Watson Clinic, Lakeland, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - South Miami Hospital, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - James A. Haley Veterans Affairs Hospital, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Memorial and Saint Elizabeth's Health Care Services LLP, Swansea, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - IU Health West Hospital, Avon, Indiana
  - IU Health Bloomington, Bloomington, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - IU Health Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Finley Hospital, Dubuque, Iowa
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Upper Chesapeake Medical Center, Bel Air, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - Tate Cancer Center, Glen Burnie, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Berkshire Hematology Oncology PC, Pittsfield, Massachusetts
  - Beth Israel Deaconess Hospital-Plymouth, Plymouth, Massachusetts
  - D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Vincent Hospital/Reliant Medical Group, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Veteran's Administration Medical Center - Ann Arbor, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren-Bay Region, Bay City, Michigan
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Huron Valley-Sinai Hospital, Commerce, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Botsford General Hospital, Farmington, Michigan
  - 21st Century Oncology-Farmington Hills, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren-Flint, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Great Lakes Cancer Institute-Lapeer Campus, Lapeer, Michigan
  - McLaren-Macomb, Mount Clemens, Michigan
  - McLaren-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - Northern Michigan Regional Hospital, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Crittenton Hospital, Rochester, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Downriver Center for Oncology, Trenton, Michigan
  - 21st Century Oncology-Troy, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center - Saint Peters, City of Saint Peters, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Kansas City Cancer Center - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Concord Hospital, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Ocean Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Princeton Radiation Oncology Center, Monroe, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Medical Center At Princeton, Princeton, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Prostate Cancer Center of New Jersey, West Orange, New Jersey
  - Lovelace Medical Center-Downtown, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Radiation Oncology Associates, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - Saint Peters Hospital-Albany, Albany, New York
  - Southside Hospital, Bay Shore, New York
  - Lourdes Hospital, Binghamton, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Veteran Affairs New York Harbor Healthcare System-Brooklyn Campus, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sands Cancer Center, Canandaigua, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore-LIJ Health System NCORP, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Highland Hospital, Rochester, New York
  - University Radiation Oncology, Rochester, New York
  - University of Rochester, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - The Coleman Radiation Center-Carteret General Hospital, Morehead City, North Carolina
  - CarolinaEast Health System-Medical Center, New Bern, North Carolina
  - Duke Cancer Institute Macon Pond, Raleigh, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - South Atlantic Radiation Oncology, Supply, North Carolina
  - Coastal Carolina Radiation Oncology, Wilmington, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Southeast Cancer Consortium-Upstate NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geaugra Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Center at Lake Medina, Medina, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Robinson Radiation Oncology, Ravenna, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Ireland Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic Wooster Specialty Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Asante Health System, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - The Regional Cancer Center, Erie, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Academic Urology Prostate Center, King of Prussia, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Upper Delaware Valley Cancer Center, Milford, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Blount Memorial Hospital, Maryville, Tennessee
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Texas Cancer Center - Medical City Dallas, Dallas, Texas
  - Texas Oncology Methodist Charlton Cancer Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - The Klabzuba Cancer Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Texas Oncology - Lewisville, Lewisville, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Texas Oncology-Wichita Falls Texoma Cancer Center, Wichita Falls, Texas
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Rutland Regional Medical Center, Rutland, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Augusta Health Cancer Center, Fishersville, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Rockingham Memorial Hospital Hahn Cancer Center, Harrisonburg, Virginia
  - Sentara Hospitals, Norfolk, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Appleton Medical Center, Appleton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin
  - Door County Cancer Center, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - The Alyce and Elmore Kraemer Cancer Care Center, West Bend, Wisconsin
  - Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (19):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA-Vancouver Island Cancer Centre, Victoria, British Columbia
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - QEII Health Sciences Centre/Capital District Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute-General Division, Ottawa, Ontario
  - Irving Greenberg Family Cancer Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Krauss DJ, Karrison T, Martinez AA, Morton G, Yan D, Bruner DW, Movsas B, Elshaikh M, Citrin D, Hershatter B, Michalski JM, Efstathiou JA, Currey A, Kavadi VS, Cury FL, Lock M, Raben A, Seaward SA, El-Gayed A, Rodgers JP, Sandler HM. Dose-Escalated Radiotherapy Alone or in Combination With Short-Term Androgen Deprivation for Intermediate-Risk Prostate Cancer: Results of a Phase III Multi-Institutional Trial. J Clin Oncol. 2023 Jun 10;41(17):3203-3216. doi: 10.1200/JCO.22.02390. Epub 2023 Apr 27. PMID 37104748

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose-Escalated Radiation Therapy Alone: Radiation therapy consists of 79.2 Gy external beam radiotherapy (EBRT) only or 45 Gy EBRT followed by low dose rate (LDR) or high-dose rate (HDR) brachytherapy. EBRT is delivered in 1.8 Gy daily fractions.
Period: Overall Study
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Started | 771 | 767
Eligible | 750 | 742
Eligible, Started Protocol Treatment, Has Adverse Event Data | 733 | 725
Eligible With Radiation Treatment Data | 725 | 707
Eligible and Consented to Quality of Life Component | 215 | 205
Completed | 750 | 742
Not Completed | 21 | 25
Not completed — Protocol Violation | 21 | 25

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation: Radiation therapy consists of 79.2 Gy EBRT only or 45 Gy EBRT followed by low- or high-dose rate brachytherapy. EBRT is delivered in 1.8 Gy daily fractions.
  Six months of androgen-deprivation therapy starts 8 weeks prior to start of radiation therapy and consists of LHRH agonist (antagonist) therapy (leuprolide, goserelin, buserelin. triptorelin, or degarelix) and anti-androgen therapy (bicalutamide or flutamide).
- Total: Total of all reporting groups
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation | Total
Number analyzed (Participants) | 750 | 742 | 1492
Age, Customized [Count of Participants; unit: Participants]
  Age: ≤ 49 years | 9 | 10 | 19
  Age: 50-59 years | 105 | 96 | 201
  Age: 60 - 69 years | 361 | 320 | 681
  Age: ≥ 70 years | 275 | 316 | 591
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 750 | 742 | 1492
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 37 | 78
  Not Hispanic or Latino | 681 | 682 | 1363
  Unknown or Not Reported | 28 | 23 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 11 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 158 | 156 | 314
  White | 557 | 554 | 1111
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 18 | 18 | 36
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 642 | 645 | 1287
    1 | 108 | 96 | 204
    Missing | 0 | 1 | 1
Number of risk factors [Count of Participants; unit: Participants] — Risk factors are defined as Gleason Score 7; 10< baseline PSA ≤20; T-Stage T2b-T2c.
  Participants
    One | 504 | 490 | 994
    Two or three | 246 | 252 | 498
Comorbidity Status [Adult Comorbidity Evaluation 27 (ACE-27) ] [Count of Participants; unit: Participants] — The Adult Comorbidity Evaluation 27 (ACE-27) is a chart-based comorbidity index providing a score (0-3) based on the number and severity of medical comorbidities for patients with cancer: 0=none, 1=mild, 2=moderate, 3=severe.
  Participants
    ACE-27 < grade 2 | 246 | 246 | 492
    ACE-27 ≥ grade 2 | 504 | 496 | 1000
Radiation Therapy Modality [Count of Participants; unit: Participants]
  Dose-escalated EBRT | 665 | 656 | 1321
  EBRT + LDR brachytherapy boost | 73 | 75 | 148
  EBRT + HDR brachytherapy boost | 12 | 11 | 23
Prostate-Specific Antigen (PSA) ng/mL [Count of Participants; unit: Participants] — Prostate-specific antigen (PSA) is a protein made by the prostate gland and found in the blood. PSA blood levels may be higher than normal in men who have prostate cancer, benign prostatic hyperplasia (BPH), or infection or inflammation of the prostate gland, and are often used to monitor patients who have been treated for prostate cancer to see if their cancer has recurred.
  Participants
    <10 | 538 | 530 | 1068
    10-20 | 212 | 212 | 424
Gleason Score [Count of Participants; unit: Participants] — Gleason score describes prostate cancer based on how abnormal the cancer cells in a biopsy sample look under a microscope. Cells are scored 1-5 with 1 indicating "low-grade" looking similar to normal cells and 5 indicating "high-grade" barely resembling normal cells due to mutation. A pathologist assigns a Gleason grade to the first and second most predominant patterns in the biopsy. The two grades are added together to calculate the Gleason score (between 2 and 10). Cancers with lower scores tend to be less aggressive, while cancers with higher scores end to be more aggressive.
  Participants
    2-6 | 64 | 59 | 123
    7 | 686 | 683 | 1369
T-Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 6th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  Participants
    T1 | 493 | 449 | 942
    T2 | 257 | 293 | 550
N-Stage [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 6th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. N0 means lymph nodes aren't involved. A higher number means the cancer is in more lymph nodes, farther away from the original tumor. NX means the lymph nodes cannot be assessed.
  Participants
    N0 | 611 | 604 | 1215
    N1 | 3 | 4 | 7
    NX | 136 | 134 | 270
M-Stage [Count of Participants; unit: Participants] — Metastasis stage per the American Joint Committee on Cancer (AJCC) 6th ed. refers to the spread of the cancer to organs and tissues in other parts of the body. M0 = No distant metastasis; M1 = Distant metastasis; MX = Distant metastasis cannot be assessed.
  Participants
    M0 | 657 | 666 | 1323
    M1 | 2 | 0 | 2
    MX | 91 | 76 | 167

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive (Overall Survival)
Description: Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided here. Analysis was planned to occur after 218 deaths were reported.
Time Frame: From randomization to last follow-up. Follow-up schedule: end of RT (2nd arm only), then every 3 months for a year, every 4 months for 4 years, then yearly. Maximum follow-up at time of analysis was 10.3 years. Five-year rates reported here.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 750 | 742
percentage of participants | 90.0 [87.7 to 92.2] | 91.0 [88.8 to 93.1]
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; This study was designed to detect an improvement in the 5-year overall survival rate from 90% (radiation alone arm) to 93.3% (radiation and androgen deprivation arm). Assuming an exponential survival distribution for each arm, this translates to a 34% relative reduction (hazard ratio 0.66) in the yearly death rate. At least 218 deaths provide 85% power with a 1-sided significance level of 0.025 and 85% power; Test type: Superiority; p = 0.22, Log Rank — One-sided significance level 0.025 (reported p-value is two-sided); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.65 to 1.11] — Reference level = radiation therapy alone arm

2. Secondary Outcome: Percentage of Participants With Biochemical Failure
Description: Biochemical failure is defined as an increase of at least 2 ng/ml above the nadir PSA. Failure time is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided here. Analysis was planned to occur after 218 deaths were reported.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 750 | 742
percentage of participants | 13.9 [11.5 to 16.6] | 7.7 [5.9 to 9.9]
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cause-specific hazard model; Test type: Superiority; p < 0.001, Log Rank — One-sided significance level 0.025 (reported p-value is two-sided); Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.39 to 0.70] — Reference level = radiation therapy alone arm
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cumulative incidence model; Test type: Superiority; p < 0.001, Gray's test — One-sided significance level 0.025 (reported p-value is two-sided)

3. Secondary Outcome: Percentage of Participants With Local Recurrence
Description: Local recurrence (failure) is defined as clinical (palpable) suspicion of local recurrence [this date is used] confirmed by biopsy. Failure time is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided here. Analysis was planned to occur after 218 deaths were reported.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 750 | 742
percentage of participants | 2.6 [1.6 to 4.1] | 0.6 [0.2 to 1.5]
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cause-specific hazard model; Test type: Superiority; p = 0.020, Log Rank — One-sided significance level 0.025 (reported p-value is two-sided); Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.22 to 0.90] — Reference level = radiation therapy alone arm
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Test type: Superiority — Cumulative incidence model; p = 0.021, Gray's test — One-sided significance level 0.025 (reported p-value is two-sided)

4. Secondary Outcome: Percentage of Participants With Regional Recurrence
Description: Regional recurrence is defined as the documented progression in pelvic lymph nodes. If discovered on image of the pelvis prompted by a biochemical failure, then the event date would be the date of documented biochemical failure.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 10.3 years.
Population: Regional recurrence data was not collected and therefore cannot be reported.
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Distant Metastasis
Description: Distant metastasis (failure) is defined as metastatic disease documented by any method. If diagnosed on diagnostic imaging prompted by biochemical failure, then the event date will be the date of biochemical progression.
  Failure time is defined as time from randomization to the date of first failure, last known follow-up (competing risk), or death without failure (censored). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided here. Analysis was planned to occur after 218 deaths were reported.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 750 | 742
percentage of participants | 3.1 [2.0 to 4.6] | 0.6 [0.2 to 1.4]
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cause-specific hazard model; Test type: Superiority; p < 0.001, Log Rank — One-sided significance level 0.025 (reported p-value is two-sided); Hazard Ratio (HR) = 0.25, 95% CI 2-sided [0.11 to 0.57] — Reference level = radiation therapy alone arm
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cumulative incidence model; Test type: Superiority; p < 0.001, Gray's test — One-sided significance level 0.025 (reported p-value is two-sided)

6. Secondary Outcome: Percentage of Participants Dead Due to Prostate Cancer (Prostate Cancer-specific Mortality)
Description: Prostate cancer specific mortality (failure) is defined as death due to prostate cancer or a complication from treatment. Failure time is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided here. Analysis was planned to occur after 218 deaths were reported.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 750 | 742
percentage of participants | 0.90 [0.4 to 1.9] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cause-specific hazard model; Test type: Superiority; p = 0.0073, Log Rank — One-sided significance level 0.025 (reported p-value is two-sided); Hazard Ratio (HR) = 0.10, 95% CI 2-sided [0.01 to 0.80] — Reference level = radiation therapy alone arm
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cumulative incidence model; Test type: Superiority; p = 0.007, Gray's test — One-sided significance level 0.025 (reported p-value is two-sided)

7. Secondary Outcome: Percentage of Participants Dead Due to Cause Other Than Prostate Cancer (Non-Prostate Cancer-specific Mortality)
Description: Non-prostate cancer specific mortality is defined as a death without evidence of prostate cancer or a complication from treatment. . Failure time is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided here. Analysis was planned to occur after 218 deaths were reported.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 750 | 742
percentage of participants | 9.1 [7.1 to 11.5] | 9.0 [7.0 to 11.4]
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cause-specific hazard model; Test type: Superiority; p = 0.52, Log Rank — One-sided significance level 0.025 (reported p-value is two-sided); Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.70 to 1.20] — Reference level = radiation therapy alone arm
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cumulative incidence model; Test type: Superiority; p = 0.56, Gray's test — One-sided significance level 0.025 (reported p-value is two-sided)

8. Secondary Outcome: Percentage of Participants Receiving Salvage Androgen Deprivation Therapy (ADT)
Description: Salvage (non-protocol) ADT administration is defined as the first administration of subsequent ADT (either LHRH agonist or anti-androgen) Failure time is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Salvage ADT rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of salvage ADT times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided here. Analysis was planned to occur after 218 deaths were reported.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 750 | 742
percentage of participants | 6.1 [4.5 to 8.1] | 4.2 [2.8 to 5.8]
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cause-specific hazard model; Test type: Superiority; p = 0.025, Log Rank — One-sided significance level 0.025 (reported p-value is two-sided); Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.41 to 0.95] — Reference level = radiation therapy alone arm
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cumulative incidence model; Test type: Superiority; p = 0.025, Gray's test — One-sided significance level 0.025 (reported p-value is two-sided)

9. Secondary Outcome: Percentage of Participants Alive (Overall Survival) by Radiation Therapy Modality
Description: Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. Five-year rates are provided here. Analysis was planned to occur after 218 deaths were reported.
Time Frame: as for outcome 1
Population: Eligible participants with radiation treatment data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 725 | 707
percentage of participants
  EBRT: number analyzed (Participants) | 645 | 623
  EBRT | 89.4 [86.9 to 91.9] | 90.3 [87.9 to 92.8]
  EBRT +LDR Brachytherapy Boost: number analyzed (Participants) | 68 | 73
  EBRT +LDR Brachytherapy Boost | 100 [100 to 100] | 97.2 [93.3 to 100.0]
  EBRT +HDR Brachytherapy Boost: number analyzed (Participants) | 12 | 11
  EBRT +HDR Brachytherapy Boost | 91.7 [76.0 to 100] | 100 [100 to 100]

10. Secondary Outcome: Number of Participants With Acute Adverse Events
Description: Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data. Acute adverse events are defined as occuring within 30 days of completion of radiation therapy.
Time Frame: From randomization to last follow-up. Follow-up schedule: end of RT (2nd arm only), then every 3 months for a year, every 4 months for 4 years, then yearly. Maximum follow-up at time of analysis was 10.3 years.
Population: Eligible participants who started protocol treatment and have adverse event data
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 733 | 725
Participants | 152 | 504
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Test type: Superiority; p < 0.001, t-test, 2 sided

11. Secondary Outcome: Percentage of Participants With Late Grade 3+ Adverse Events
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data. Late adverse events are defined as occurring more than 30 days after the end of radiation therapy. Failure is defined as grade 3 or higher late adverse event. Failure time is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided here. Analysis was planned to occur after 218 deaths were reported.
Time Frame: From randomization to last follow-up. Follow-up schedule: end of RT (2nd arm only), then every 3 months for a year, every 4 months for 4 years, then yearly. Maximum follow-up at time of analysis was 10.3 years. Five-year rates are reported here.
Population: Eligible participants who started protocol treatment and have adverse event data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 733 | 725
percentage of participants | 12.8 [10.5 to 15.4] | 15.2 [12.6 to 17.9]
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Test type: Superiority; p = 0.13, Gray's test — One-sided significance level 0.025 (reported p-value is one-sided); Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.89 to 1.53] — Reference level = radiation therapy alone arm

12. Secondary Outcome: Percentage of Participants Failed (Freedom From Failure)
Description: Failure is defined as biochemical failure, local failure, or distant metastasis. Failure time is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Five-year rates are provided here. Analysis was planned to occur after 218 deaths were reported.
Time Frame: as for outcome 11
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 750 | 742
percentage of participants | 14.8 [12.2 to 17.5] | 7.9 [6.0 to 10.1]
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cause-specific hazard model; Test type: Superiority; p < 0.001, Log Rank — One-sided significance level 0.025 (reported p-value is two-sided); Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.39 to 0.70] — Reference level = radiation therapy alone arm
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Cumulative incidence model; Test type: Superiority; p < 0.001, Gray's test — One-sided significance level 0.025 (reported p-value is two-sided)

13. Secondary Outcome: Change From Baseline in Expanded Prostate Cancer Index Composite (EPIC) Urinary Domain Score
Description: The EPIC assesses disease-specific aspects of prostate cancer and it's therapies and consists of four summary domains (bowel, urinary, sexual, and hormonal), each ranging from 0-100, with higher scores representing better health-related quality of life. Change is calculated as time point value - baseline value, such that a positive change indicates improvement.
Time Frame: Last week of RT (approximately 9 and 17 weeks from start of protocol treatment for Arm 1 and 2, respectively), then 6 months, 1 year and 5 years from end of RT.
Population: Eligible participants who consented to quality of life component and have data at baseline and time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Dose-Escalated Radiation Therapy Alone (Arm 1): Radiation therapy consists of 79.2 Gy EBRT only or 45 Gy EBRT followed by low- or high-dose rate brachytherapy. EBRT is delivered in 1.8 Gy daily fractions.
- Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation (Arm 2): Radiation therapy consists of 79.2 Gy EBRT only or 45 Gy EBRT followed by low- or high-dose rate brachytherapy. EBRT is delivered in 1.8 Gy daily fractions.
  Six months of androgen-deprivation therapy starts 8 weeks prior to start of radiation therapy and consists of LHRH agonist (antagonist) therapy (leuprolide, goserelin, buserelin. triptorelin, or degarelix) and anti-androgen therapy (bicalutamide or flutamide).
Arm/Group | Dose-Escalated Radiation Therapy Alone (Arm 1) | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation (Arm 2)
Number analyzed (Participants) | 215 | 205
score on a scale
  End of RT: number analyzed (Participants) | 202 | 185
  End of RT | -12.4 (17.0) | -13.8 (15.4)
  Six months post-RT: number analyzed (Participants) | 180 | 179
  Six months post-RT | -0.1 (14.9) | -3.6 (15.3)
  One year post-RT: number analyzed (Participants) | 174 | 171
  One year post-RT | -1.9 (15.9) | -1.6 (15.3)
  Five years post-RT: number analyzed (Participants) | 138 | 145
  Five years post-RT | -0.4 (14.9) | 0.3 (12.3)
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone (Arm 1) vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation (Arm 2); End of RT; Test type: Superiority; p = 0.38, t-test, 2 sided
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone (Arm 1) vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation (Arm 2); 6 months post-RT; Test type: Superiority; p = 0.032, t-test, 2 sided
Statistical Analysis 3: Comparison: Dose-Escalated Radiation Therapy Alone (Arm 1) vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation (Arm 2); One year post-RT; Test type: Superiority; p = 0.87, t-test, 2 sided
Statistical Analysis 4: Comparison: Dose-Escalated Radiation Therapy Alone (Arm 1) vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation (Arm 2); Five years post-RT; Test type: Superiority; p = 0.67, t-test, 2 sided

14. Secondary Outcome: Change From Baseline in Expanded Prostate Cancer Index Composite (EPIC) Bowel Domain Score
Description: as for outcome 13
Time Frame: as for outcome 13
Population: Eligible participants who consented to quality of life component and have data at baseline and time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 215 | 205
score on a scale
  End of RT: number analyzed (Participants) | 203 | 186
  End of RT | -9.7 (14.7) | -10.5 (13.7)
  Six months post-RT: number analyzed (Participants) | 178 | 182
  Six months post-RT | -2.6 (12.8) | -3.8 (9.6)
  One year post-RT: number analyzed (Participants) | 177 | 171
  One year post-RT | -4.0 (12.8) | -5.2 (13.4)
  Five years post-RT: number analyzed (Participants) | 137 | 145
  Five years post-RT | -2.7 (13.2) | -2.9 (10.7)
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; End of RT; Test type: Superiority; p = 0.58, t-test, 2 sided
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Six months post-RT; Test type: Superiority; p = 0.31, t-test, 2 sided
Statistical Analysis 3: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; One year post-RT; Test type: Superiority; p = 0.36, t-test, 2 sided
Statistical Analysis 4: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Five years post-RT; Test type: Superiority; p = 0.88, t-test, 2 sided

15. Secondary Outcome: Change From Baseline in Expanded Prostate Cancer Index Composite (EPIC) Hormonal Domain Score
Description: as for outcome 13
Time Frame: as for outcome 13
Population: Eligible participants who consented to quality of life component and have data at baseline and time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 215 | 205
score on a scale
  End of RT: number analyzed (Participants) | 199 | 187
  End of RT | -1.8 (10.2) | -18.4 (16.2)
  Six months post-RT: number analyzed (Participants) | 174 | 181
  Six months post-RT | -0.7 (11.9) | -13.7 (16.9)
  One year post-RT: number analyzed (Participants) | 173 | 175
  One year post-RT | -0.8 (14.7) | -7.8 (14.4)
  Five years post-RT: number analyzed (Participants) | 133 | 138
  Five years post-RT | -0.3 (15.9) | -2.7 (13.9)
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; End of RT; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Six months post-RT; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; One year post-RT; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Five years post-RT; Test type: Superiority; p = 0.18, t-test, 2 sided

16. Secondary Outcome: Change From Baseline in Expanded Prostate Cancer Index Composite (EPIC) Sexual Domain Score
Description: as for outcome 13
Time Frame: as for outcome 13
Population: Eligible participants who consented to quality of life component and have data at baseline and time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 215 | 205
score on a scale
  End of RT: number analyzed (Participants) | 189 | 180
  End of RT | -6.7 (18.9) | -22.6 (25.8)
  Six months post-RT: number analyzed (Participants) | 172 | 168
  Six months post-RT | -7.9 (23.0) | -19.9 (25.3)
  One year post-RT: number analyzed (Participants) | 173 | 165
  One year post-RT | -8.5 (22.7) | -16.6 (23.7)
  Five years post-RT: number analyzed (Participants) | 129 | 138
  Five years post-RT | -10.0 (26.6) | -9.6 (27.6)
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; End of RT; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Six months post-RT; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; One year post-RT; Test type: Superiority; p = 0.0014, t-test, 2 sided
Statistical Analysis 4: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Five years post-RT; Test type: Superiority; p = 0.90, t-test, 2 sided

17. Secondary Outcome: Change From Baseline in Patient Reported Outcome Measurement Information System (PROMIS) Fatigue Domain Score
Description: The PROMIS Fatigue short form 8a contains 8 questions, each with 5 responses ranging from 1 to 5, evaluating self-reported fatigue symptoms over the past 7 days. The total score is the sum of all questions which is then converted into a pro-rated T-score with a mean of 50 and standard deviation of 10, with a possible range of 33.1 to 77.8. Higher scores indicate more fatigue. Change is defined as value at one year - value at baseline. Positive change from baseline indicates increased fatigue at one year.
Time Frame: as for outcome 13
Population: Participants who consented to QOL component and have data at baseline and timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 215 | 205
score on a scale
  End of RT: number analyzed (Participants) | 201 | 187
  End of RT | 0.80 (4.66) | 1.84 (5.54)
  Six months post-RT: number analyzed (Participants) | 199 | 186
  Six months post-RT | 1.09 (5.14) | 1.21 (5.34)
  One year post_RT: number analyzed (Participants) | 199 | 188
  One year post_RT | 0.99 (6.00) | 0.86 (5.08)
  Five years post-RT: number analyzed (Participants) | 195 | 186
  Five years post-RT | 0.97 (6.71) | 0.80 (5.62)
Statistical Analysis 1: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; End of RT; Test type: Superiority; p = 0.046, t-test, 2 sided
Statistical Analysis 2: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; 6 months post-RT; Test type: Superiority; p = 0.82, t-test, 2 sided
Statistical Analysis 3: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; One year post-RT; Test type: Superiority; p = 0.82, t-test, 2 sided
Statistical Analysis 4: Comparison: Dose-Escalated Radiation Therapy Alone vs Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation; Five years post-RT; Test type: Superiority; p = 0.79, t-test, 2 sided

18. Secondary Outcome: Quality Adjusted Life Years (QALYs)
Time Frame: as for outcome 13
Population: The protocol states that this outcome measure will be analyzed only if the primary endpoint hypothesis is substantiated, which it was not. Therefore no patients were analyzed.
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Correlation Between PROMIS Fatigue Score Change and Plasma Cytokine Change
Time Frame: From date of randomization to 3 weeks from start of RT.
Population: The protocol did not provide sufficient detail to meet current National Cancer Institute requirements for release of specimens from the NRG Oncology tissue bank for the protocol-specified analysis, therefore no assays were performed, and no data were collected for this outcome measure (cytokine levels). Specimen use will require future federal approval and funding separate from this trial.
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: End of RT (2nd arm only), then every 3 months for a year, every 4 months for 4 years, then yearly. Maximum follow-up at time of analysis was 10.3 years.
Description: All-cause mortality was assessed in eligible participants. Adverse events were assessed in eligible participants who started protocol treatment and had adverse event data.
Arm/Group | Dose-Escalated Radiation Therapy Alone | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation
All-Cause Mortality (participants affected / at risk) | 119/750 | 100/742
Serious Adverse Events (participants affected / at risk) | 20/733 | 33/725
Other Adverse Events (participants affected / at risk) | 597/733 | 647/725
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-Escalated Radiation Therapy Alone (N=733) | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation (N=725)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 1 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 1
Cardiopulmonary arrest (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 5
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 3 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 2
Rectal pain (Gastrointestinal disorders) | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 1
Autoimmune disorder (Immune system disorders) | 1 | 0
Abdominal infection [with unknown ANC] (Infections and infestations) | 0 | 1
Bladder infection [with unknown ANC] (Infections and infestations) | 0 | 1
Bone infection [with unknown ANC] (Infections and infestations) | 0 | 1
Neck NOS infection [other] (Infections and infestations) | 1 | 0
Sepsis [with unknown ANC] (Infections and infestations) | 0 | 1
Soft tissue infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1
Soft tissue infection [with unknown ANC] (Infections and infestations) | 0 | 1
Urinary tract infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 2
Urinary tract infection [with unknown ANC] (Infections and infestations) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Cardiac troponin I increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Serum cholesterol increased (Investigations) | 0 | 1
Weight loss (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Blood glucose increased (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Serum potassium decreased (Metabolism and nutrition disorders) | 1 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1
Neurological disorder NOS (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Hemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 3 | 0
Urinary retention (Renal and urinary disorders) | 4 | 2
Urogenital disorder (Renal and urinary disorders) | 2 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-Escalated Radiation Therapy Alone (N=733) | Dose-Escalated Radiation Therapy and Short-Term Androgen-Deprivation (N=725)
Hemoglobin decreased (Blood and lymphatic system disorders) | 30 | 74
Constipation (Gastrointestinal disorders) | 86 | 96
Diarrhea (Gastrointestinal disorders) | 134 | 186
Gastrointestinal disorder (Gastrointestinal disorders) | 72 | 77
Hemorrhoids (Gastrointestinal disorders) | 43 | 47
Proctitis (Gastrointestinal disorders) | 105 | 115
Rectal hemorrhage (Gastrointestinal disorders) | 105 | 93
Fatigue (General disorders) | 210 | 338
Pain [other] (General disorders) | 37 | 49
Alanine aminotransferase increased (Investigations) | 2 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 46
Dizziness (Nervous system disorders) | 12 | 38
Libido decreased (Psychiatric disorders) | 45 | 121
Cystitis (Renal and urinary disorders) | 74 | 78
Urethral pain (Renal and urinary disorders) | 30 | 44
Urinary frequency (Renal and urinary disorders) | 462 | 531
Urinary incontinence (Renal and urinary disorders) | 125 | 136
Urinary retention (Renal and urinary disorders) | 180 | 222
Urogenital disorder (Renal and urinary disorders) | 158 | 200
Ejaculation disorder (Reproductive system and breast disorders) | 34 | 38
Erectile dysfunction (Reproductive system and breast disorders) | 273 | 359
Hot flashes (Vascular disorders) | 23 | 414

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT00936390/Prot_SAP_000.pdf
  • Informed Consent Form (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT00936390/ICF_001.pdf